CLINICAL TRIAL: NCT04898244
Title: Causes of High Caesarean Section Rates in Egypt: Perception of Obstetricians
Brief Title: Obstetricians' Views on the Reasons for Egypt's High Caesarean Section Rates
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saad El Gelany,MD, Professor, Minia University
Other Study IDs: MUEOB0022
Record Dates: First submitted 2021-05-15; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Caesarean Section Rate; Egypt
Keywords: Caesarean Section; high CS rates; Egypt; Minia university; Obstetricians

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Handling of questionnaires to a number of obstetricians from different hospitals to show their perceptions about causes of high cs rate in Egypt

DETAILED DESCRIPTION:
An open-ended self-administered questionnaire Handled to a number of obstetricians from different hospitals to show their perceptions about causes of the high cs rate in Egypt.

ELIGIBILITY:
Inclusion Criteria:

Obstetricians from different hospitals. -

Exclusion Criteria:

Refusal to participate

-

Ages: 28 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Obstetricians from different hospitals and areas
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Reasons of the High Caesarean Section Rates in Egypt. | 12 months
  A questionnaire filled by Obstetricians working in Egypt to explore the reasons of high Caesarean Section Rates from their point of view.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt